CLINICAL TRIAL: NCT02534064
Title: Effect of the Consumption of Yogurt Fortified in Calcium and Vitamin D on the Circulating Levels of 25OHD in Postmenopausal Women
Brief Title: Effect of Consumption of Yogurt Fortified in Calcium and Vit. D on Circulating Levels of 25OHD in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yoplait France SAS (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CATWIN2107
Record Dates: First submitted 2015-08-19; First posted 2015-08-27 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Menopause; Vitamin D Deficiency
Keywords: Menopause; Osteoporosis; Hip fractures; vitamin D deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis; Hip Fractures | interventions — calin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A: 2 yogurts (Experimental): consumption of 2 CALIN+ pots per day during 16 weeks and follow up without product intake during 8 weeks.
  Interventions: Dietary Supplement: CALIN+
- Group B: 1 yogurt (Experimental): consumption of 1 CALIN+ pot per day during 16 weeks and follow up without product during 8 weeks.
  Interventions: Dietary Supplement: CALIN+
- Group C: No yogurt (No Intervention): no changes in dietary habits during 24 weeks.

INTERVENTIONS:
Dietary Supplement: CALIN+ — Consumption of 2 CALIN+ pots per day during 16 weeks and follow up without product intake during 8 weeks.
  Arms: Group A: 2 yogurts
Dietary Supplement: CALIN+ — Consumption of 1 CALIN+ pot per day during 16 weeks and follow up without product intake during 8 weeks.
  Arms: Group B: 1 yogurt

SUMMARY:
The purpose of this study is to evaluate the effect of daily consumption of one or two CALIN+ pot(s) versus no intake of product, after 4, 8, 12 and 16 weeks, on the evolution of the serum concentration of 25-hydroxy vitamin D (25OHD) (D2 + D3) in postmenopausal women.

DETAILED DESCRIPTION:
The active form of vitamin D is produced by skin when it is exposed to ultraviolet-B (UVB) rays. However, because of our sedentary lifestyle and to the low sun exposure during winter, the vitamin D status is most frequently deficient. Hence the consumption of enriched food could be an efficient strategy to improve vitamin D status.

The current recommendation for vitamin D intake is 20 µg per day for adults (19-50 yo) and between 25 and 37.5 µg per day for people over 50 years old according to the French National Medicine Academy. However, the recommended daily allowance (RDA) in France for vitamin D is limited to 5 µg corresponding to the maximum enrichment allowed in a food product. The current study is designed to evaluate if a daily consumption of two CALIN+ yogurts enriched with 5µg of vitamin D is sufficient to improve the vitamin D status in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject, aged between 55 and 75 years inclusive.
2. Menopausal female subject for more than 5 years.
3. Non smoker or smoker less than 5 cigarettes a day
4. Body Mass Index (BMI) between 18 and 28 kg/m² inclusive.
5. Subject with a serum 25-hydroxyvitamin D2 + D3 between 10 and 30 ng/mL corresponding to a vitamin D insufficiency.
6. Subject with a Mini Nutritional Assessment (MNA) > 20.
7. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
8. Normal blood pressure (BP) and heart rate (HR) at the screening visit after 10 minutes in supine position:

   * 95 mmHg ≤ systolic blood pressure (SBP) ≤ 160 mmHg,
   * 50 mmHg ≤ diastolic blood pressure (DBP) ≤ 95 mmHg,
   * 40 bpm ≤ HR (heart rate) ≤ 80 bpm.
9. Subject with normal dietary habits (no vegetarian, lactose intolerant, gluten-free subject).
10. Having given a written informed consent prior to selection.
11. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. Subject who have taken any form of vitamin D supplementation in the 6 months preceding the study, including through fortified food (milk, dairy products, oil and tofu) or food supplements.
2. Subject who consumed more than 3 dairy products per day.
3. Functional impotence.
4. Concomitant bone disease or affecting mineral metabolism, in whatever form.
5. History of bone fracture in the previous year.
6. Presence of a primary hyperparathyroidism, chronic gastrointestinal disease or patent hepatic and/or renal impairment or a progressive severe disease.
7. Type 1 diabetic subject.
8. Subject with eating disorder.
9. Subject with a treatment which can interfere with the study purpose at the moment of recruitment or 6 months before (see section 5.6)
10. Significant allergies or food intolerance.
11. Subject who cannot be contacted in case of emergency.
12. History or presence of drug or alcohol abuse (alcohol consumption > 5 glasses / day).
13. Medical and surgical history which, in the judgment of the Investigator, is not compatible with this study.
14. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, or has poor mental development.
15. Blood donation within two months before the study beginning.
16. Subject in the exclusion period of a previous study or subject who refuse to be on the "Fichier National des Volontaires Sains".
17. Subject who refuse to sign the Informed Consent Form.
18. Participation to another study within 3 months prior the study beginning.
19. Subject under administrative or legal supervision.
20. Subject who are deprived of their liberty by judicial of administration decision.
21. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change of serum 25OHD (D2 + D3) concentration over the 16 weeks | serum 25OHD (D2 + D3) concentration will be evaluated at 4, 8, 12 and 16 weeks

SECONDARY OUTCOMES:
Serum ParaThyroid Hormone (PTH) level | Evolution after 16 weeks consumption period
  Serum (ParaThyroid Hormone) PTH level
Serum calcium level | Evolution after 16 weeks consumption period
  Serum calcium level
Serum 25OHD (D2 + D3) level | Evolution after 16 weeks consumption period
  Serum 25OHD (D2 + D3) level
Diastolic / systolic blood pressures (mm/Hg) | Evolution after 16 weeks consumption period
  Diastolic / systolic blood pressures
Weight (kg) | Evolution after 16 weeks consumption period
  Weight (kg)
Waist circumference (cm) | Evolution after 16 weeks consumption period
  Waist circumference (com)
Rate constant | over two months
  Rate constant
Serum 25OHD (D2 + D3) level | Evolution over 8 weeks consumption period for women included in study during winter (before March 1, 2015)
  Serum 25OHD (D2 + D3) level
Serum ParaThyroid Hormone (PTH) level | Evolution over 8 weeks consumption period for women included in study during winter (before March 1, 2015)
  Serum ParaThyroid Hormone (PTH) level
Serum calcium level | Evolution over 8 weeks consumption period for women included in study during winter (before March 1, 2015)
  Serum calcium level
Diastolic/systolic blood pressures (mm/Hg) | Evolution over 8 weeks consumption period for women included in study during winter (before March 1, 2015)
  Diastolic/systolic blood pressures (mm/Hg)
Weight (kg) | Evolution over 8 weeks consumption period for women included in study during winter (before March 1, 2015)
  Weight (kg)
Waist circumference (cm) | Evolution over 8 weeks consumption period for women included in study during winter (before March 1, 2015)
  Waist circumference (cm)
Serum levels of 25OHD (D2 + D3), | Evolution over the 2 months follow up period
  Serum levels of 25OHD (D2 + D3),
Serum ParaThyroid Hormone (PTH) level | Evolution over the 2 months follow up period
  Serum ParaThyroid Hormone (PTH) level
Assessment of sun exposure and dietary vitamin D intake using the Garabedian questionnaire | 4 months and 6 months
  Assessment of sun exposure and dietary vitamin D intake using the Garabedian questionnaire
Assessment of calcium intake using a simplified calcium questionnaire | over the 16-week consumption period and over the first 8 weeks consumption for women included in the study during the winter season, i.e. before March 1, 2015.
  Assessment of calcium intake using a simplified calcium questionnaire
Compliance of CALIN+ consumption reported in diary | up to 20 weeks
  Number of consumed yogurt per day
Acceptability of CALIN+ consumption by questionnaire | up to 20 weeks
  Change from baseline in acceptability score (0: do not agree at all; 10: agree completely)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Latreille-Barbier, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France